CLINICAL TRIAL: NCT06159309
Title: Quality of Life After Hyperbaric Oxygen Therapy in Post-COVID Patients
Acronym: QoL COVID HBOT
Status: Active, not recruiting | Type: Observational
Sponsor: Rutger Lalieu (Other)
Responsible Party: Sponsor-Investigator, Rutger Lalieu, Principal Investigator, Hyperbaar Geneeskundig Centrum Rijswijk
Organization: Hyperbaar Geneeskundig Centrum Rijswijk (Other)
Other Study IDs: MEC-2023-0433
Record Dates: First submitted 2023-12-04; First posted 2023-12-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Long COVID; Long COVID-19 Syndrome; Long Covid19; Long Covid 19
Keywords: registry; covid; long-covid; post-covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long Covid patients: All post-COVID patients that are referred for hyperbaric oxygen (and that are eligible for treatment)
  Interventions: Other: Hyperbaric oxygen therapy

INTERVENTIONS:
Other: Hyperbaric oxygen therapy — HBOT per local protocol, i.e. 40 sessions 2.4 ATA, at the discretion of the hyperbaric physician

SUMMARY:
Post-Covid syndrome, also known as long Covid, is a clinical condition in which patients experience long term symptoms after Covid-19 infection. Treatment options for post-Covid are not effective. Therefore, there is an urgent need for a novel therapy. The first study results of HBOT in post-Covid patients are promising. Previous research from Israel has shown improvements in quality of life after HBOT. However, long term results are unknown. Therefore, this study aims to evaluate quality of life at one year after hyperbaric oxygen therapy in post-Covid patients with cognitive symptoms. It is hypothesized that quality of life at one year after HBOT is improved. Furthermore, this study aims to evaluate return to work after HBOT. To our knowledge this was not done before. An observational prospective cohort study will be conducted to answer the research questions. All post-Covid patients who are treated with hyperbaric oxygen therapy in participating centers, will be eligible for inclusion. Questionnaires and medical doctor consultations will be used in order to collect all data.

There are no risks for participants, since only 7 questionnaires are not part of standard clinical care. The burden is approximately 40 minutes extra in total for participants, compared to standard clinical care.

DETAILED DESCRIPTION:
The study design is a prospective observational cohort study. Questionnaires and medical doctor consultations will be used in order to collect all data. All patients treated with HBOT have medical doctor consultations at baseline and every 10th session of HBOT (standard clinical care).

At baseline, the following characteristics will be collected: gender, age, BMI, medical history, Covid infection information, vaccination status, work status before Covid infection, previous Covid treatments, hospital and/or intensive care unit admission during Covid infection and smoking status. Furthermore, all patients treated are asked to fill out the SF-36 and EQ-5D questionnaires, a proprietary post-Covid symptoms questionnaire, and a questionnaire regaring work status. These questionnaires are repeated after 20, 40 (50) sessions of HBOT and after 3 and 12 months after the last treatment session.

During the following medical doctor consultations, side effects, changes in medication and interruptions of HBOT will be recorded as well to monitor compliance.

An interim analysis will be performed after 6 months to continue or stop treatments, based on the clinical results (as measured with the Physical Component Score of the SF-36 questionnaire). The minimal clinically important difference (MCID) to warrant early termination of therapy is if <5% of patients improves 3 points. The upper limit (and reason to continue) is if >50% achieve an MCID of 7 points.

ELIGIBILITY:
Inclusion Criteria:

* Long COVID patients who are reffered for treatment with hyperbaric oxygen therapy
* Patients are suffering from cognitive symptoms for >3 months after Covid infection

Exclusion Criteria:

* Patients who are not able to fill in questionnaires and informed consent.
* Patients who can't read or do not understand the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will consist of post-Covid patients from the Netherlands, who are treated with hyperbaric oxygen therapy at several different treatment centers. All patients are adults and will receive standard clinical hyperbaric oxygen therapy at these clinics.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Quality of life 3 and 12 months | 3 and 12 months
  Is the expected improvement in quality of life in Long COVID patients after treatment with HBOT maintained at 12-months follow-up

SECONDARY OUTCOMES:
Long Covid symptoms | 3 and 12 months
  What symptoms do Long COVID patients who were referred for HBOT suffer from?
Cognitive complaints | 3 and 12 months
  Is there any improvement of symptoms in Long COVID patients with cognitive symptoms during HBOT and after HBOT?
Work | 3 and 12 months
  Do changes in absence at work occur after treatment with HBOT in Long COVID patients with cognitive symptoms?
Risk factors quality of life | 3 and 12 months
  What are risk factors for low health related quality of life in Long COVID patients with cognitive symptoms who are treated with HBOT?
Profile of non-responders versus responders | 3 and 12 months
  What are the differences in baseline characteristics of patients that are non-responders and responders after HBOT?

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - DVK Hogeveen, Hoogeveen, Drenthe
  - DVK Geldrop, Geldrop, North Brabant
  - DVK Waalwijk, Waalwijk, North Brabant
  - HGC Rijswijk, Rijswijk, South Holland
  - DVK Rotterdam, Rotterdam, South Holland
  - DVK Amersfoort, Amersfoort, Utrecht

IPD SHARING:
Plan to Share IPD: No
The data is retrieved from patient files (after informed consent). Even though the data is pseudonymised, there is too much risk of confidentialty breach.